CLINICAL TRIAL: NCT03758651
Title: Williams Syndrome SHAAPE STUDY [Strength, Hormones, Activity & Adiposity, DNA Programming, Eating Study]
Brief Title: Williams Syndrome Strength, Hormones, Activity & Adiposity, DNA Programming, Eating Study
Acronym: SHAAPE
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Williams Syndrome Association (Unknown)
Responsible Party: Principal Investigator, Barbara R. Pober, Geneticist, MGH and Professor of Pediatrics (Emeritus), Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2018P000633
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Williams Syndrome; Lipedema
Keywords: Williams Syndrome; Lipedema; Body Composition; Glucose; Bone Density
MeSH Terms: conditions — Williams Syndrome; Lipedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Williams syndrome - Onsite participation: Individuals with Williams syndrome who will participate in the study at Massachusetts General Hospital (MGH)
- Williams syndrome - Convention participation: Individuals with Williams syndrome (WS) who will have a more limited evaluation at a convention focusing on WS, such as the WS Association convention.
- Williams syndrome - Remote participation: Individuals with Williams syndrome (WS) who will participate in the study remotely by filling out a questionnaire and providing information by mail.
- Healthy Controls: Healthy individuals without Williams syndrome who will participate in the study at the Massachusetts General Hospital

SUMMARY:
Williams syndrome (WS) is a rare microdeletion genetic disorder that has a broad phenotype including many endocrine and metabolic abnormalities. Dr. Pober and colleagues at MGH have reported the following findings in adults with WS: abnormal body composition (excess body fat accumulation with a lipedema phenotype), decreased bone mineral density, abnormal glucose tolerance, and reduced lean mass. Despite the high prevalence and potential effect of metabolic abnormalities on the health of persons with WS, their full phenotypic range, potential causal factors (either genetic and/or hormonal) along with their impact on other aspects of health (such as risk of falls and fractures or interaction with emotional behavioral concerns) remain incompletely characterized. The purpose of the current study in a large cohort of subjects with WS is to: collect further information to characterize the timing of onset and distribution of body fat; better characterize hormonal status of WS subjects; and screen for genetic variation using single-nucleotide-polymorphism (SNP) analysis that could elucidate genetic contributors to the lipedema phenotype as well as the other observed metabolic and bone abnormalities.

ELIGIBILITY:
For those participating in-person at Massachusetts General Hospital:

Inclusion Criteria

1. Male or Female age 18-70 years old
2. Diagnosis of Williams syndrome (WS), established by experienced clinician, parent report, or confirmed by genetic testing such as FISH (fluorescent in situ hybridization) or chromosomal microarray (WS only)
3. Availability of a parent or guardian to review details of the study with their family member with WS and participate in the consent process (all WS regardless of age)
4. Availability of a parent or guardian to provide selected medical information (WS only)

Exclusion Criteria

1. History of weight loss surgery or liposuction
2. Positive urine pregnancy test (females only)
3. Obesity or abnormal fat distribution due to a known secondary cause (except WS) such as Cushing syndrome, HIV-infection, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dr. Pober and colleagues plan to include 30 individuals with Williams syndrome (WS) who participate at Massachusetts General Hospital, along with 25-30 matched control individuals, as well as 50 individuals with WS who participate at conventions related to WS, and 100 individuals with WS who participate remotely.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density - Lumbar Spine | baseline only
Whole Body DEXA (dual energy x-ray absorptiometry) scan | baseline only
  To assess body proportions of fat, bone, and muscle

SECONDARY OUTCOMES:
Bone Mineral Density - Hip | baseline only
Resting energy expenditure | baseline only
Serum Total Testosterone | baseline only
Serum Estrogen | baseline only
Fasting blood sugar and Oral glucose tolerance test (OGTT) | baseline only

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited and de-identified dataset may be available to other researchers at the conclusion of the study.